CLINICAL TRIAL: NCT01820754
Title: Evaluation of Circulating T Cells and Tumor Infiltrating Lymphocytes With Specificities Against Tumor Associated Antigens During and After Neoadjuvant Chemotherapy and Phased Ipilimumab in Non-Small Cell Lung Cancer
Brief Title: Evaluation of Circulating T Cells and Tumor Infiltrating Lymphocytes (TILs) During / After Pre-Surgery Chemotherapy in Non-Small Cell Lung Cancer (NSCLC)
Acronym: TOP1201 IPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00038093
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Lung Cancer; Non Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Ipilimumab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab (Experimental): Neoadjuvant (Pre-Surgery): Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes Adjuvant (Post-Surgery): Ipilimumab 10 mg/kg IV every 3 weeks times 2 doses beginning 4 weeks postoperative ( up to 10 weeks if needed for recovery) Maintenance: Ipilimumab 10 mg/kg/IV every 12 weeks times 2 doses
  Interventions: Drug: Ipilimumab; Drug: Paclitaxel, Cisplatin, Carboplatin

INTERVENTIONS:
Drug: Ipilimumab — Neoadjuvant (Pre-Surgery): Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes
  Adjuvant (Post-Surgery): Ipilimumab 10 mg/kg IV every 3 weeks times 2 doses beginning 4 weeks postoperative ( up to 10 weeks if needed for recovery)
  Maintenance: Ipilimumab 10 mg/kg/IV every 12 weeks times 2 doses
  Other Names: Yervoy
Drug: Paclitaxel, Cisplatin, Carboplatin — Neoadjuvant (Pre-Surgery) Cycle 1: Paclitaxel 175 mg/m2 IV over 3 hours , followed by Cisplatin 75 mg/m2 IV over 60 minutes or carboplatin AUC 6 IV over 30-60 minutes on day 1(Every 21 days x 1 cycle)
  Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes, Paclitaxel 175 mg/m2 IV over 3 hours , followed by Cisplatin 75 mg/m2 IV over 60 minutes or carboplatin AUC 6 IV over 30-60 minutes on day 1(Every 21 days x 2 cycles)
  Other Names: Taxol, Platinol, Paraplatin

SUMMARY:
The purpose of this study is to evaluate whether the combination of neoadjuvant chemotherapy (chemotherapy before surgery) plus ipilimumab for lung cancer increases the number of patients with detectable circulating T cells with specificities against tumor associated antigens (TAA) from zero percent (0%) of patients prior to therapy to 20% of patients after neoadjuvant chemotherapy plus ipilimumab.

This is an open label Phase 2 trial. Patients with clinical stage 1B (>4 cm), 2, (N0-2) or 3 non-small cell lung cancer (NSCLC) and no prior therapy for the current diagnosis of lung cancer will be eligible for the study. Subjects will receive 3 cycles of neoadjuvant chemotherapy (paclitaxel + cisplatin/carboplatin). Ipilimumab will be administered during Cycles 2 and 3 of standard chemotherapy and for up to 4 cycles alone after surgery. Subjects will undergo standard clinically indicated surgical resection of their lung cancer as deemed appropriate by their surgeon.

Standard diagnostic and staging work up will be performed including: pathologic/histologic diagnosis of NSCLC, Positron Emission Tomography (PET)/Computed Tomography (CT) scan, brain imaging, and mediastinoscopy. Three cycles of neoadjuvant chemotherapy will be given. Ipilimumab will be added to neoadjuvant chemotherapy for cycles 2 and 3. Standard surgical evaluation and therapy will be performed following completion of neoadjuvant therapy. Two cycles of single agent ipilimumab will be given after surgery (adjuvantly), followed by 2 cycles of maintenance therapy.

DETAILED DESCRIPTION:
The investigators propose studying the cell mediated effects of ipilimumab in combination with chemotherapy in the neoadjuvant setting for NSCLC. The overall immune assessment strategy for the proposed ipilimumab neoadjuvant trial will be based on the hypothesis that 1) T cells with specificities against tumor associated antigens expressed by the patient's progressing NSCLC are present, but functionally impaired, at baseline, and 2) that the immunomodulatory effects of chemotherapy plus ipilimumab will impact the suppressive mechanisms, restoring functional reactivity to important anti-tumor effector cell populations.

An important potential biomarker for anti-tumor immune response is the proliferation and stimulation of circulating T cells with specificities against tumor associated antigens (TAA). At baseline few patients with cancer have populations of circulating T cells with specificities against TAA above the detectable level of 0.05% CD8 lymphocytes. The primary endpoint of this clinical trial will be to determine if the addition of ipilimumab to neoadjuvant chemotherapy for non-small cell lung cancer increases the percentage of patients with circulating T cells with specificities against TAA. We will also measure tumor infiltrating lymphocytes in resected tumors.

Study Interventions:

The investigational agent, ipilimumab, will be added to neoadjuvant chemotherapy for cycles 2 and 3. Standard surgical evaluation and therapy will be performed following completion of neoadjuvant therapy. Two cycles of single agent ipilimumab will be given after surgery (adjuvantly), followed by 2 cycles of maintenance therapy.

Neoadjuvant:

Cycle 1: Paclitaxel 175 mg/m2 IV over 3 hours followed by cisplatin 75 mg/m2 over 60 minutes or carboplatin Area Under Curve (AUC) 6 (capped at 900 mg)over 30-60 minutes on day 1 (every 21 days x 1 cycle) Cycles 2 and 3: Ipilimumab 10mg/kg IV over 90 minutes, Paclitaxel 175 mg/m2 over 3 hours followed by cisplatin 75 mg/m2 or carboplatin AUC 6 (capped at 900 mg)IV over 30-60 minutes (every 21 days x 2 cycles) Surgery: Standard surgical evaluation will occur at least 21 days after the last dose (Cycle 3) of chemotherapy followed by surgical therapy.

Post-surgical Therapy: (Total of 4 doses of ipilimumab will be given post-operatively):

Adjuvant: Ipilimumab 10 mg/kg IV every 3 weeks x 2 doses, beginning 4 weeks postoperative (up to 10 weeks if needed for recovery) Maintenance: Ipilimumab 10 mg/kg IV every 12 weeks x 2 doses

Correlative Science Measures: Study specific research blood and tissue test(s) will be conducted:

Blood Specimens:

•Peripheral blood mononuclear cells (PBMC) isolated from freshly drawn anti-coagulated blood will be analyzed for circulating T cells with specificities against tumor-associated antigens (TAA) at 4 time points, namely 1) Baseline prior to treatment, 2) cycle 2, prior to ipilimumab therapy, 3) 21-36 days after completion of cycle 3 chemotherapy prior to surgery, and 4) 3-6 weeks after adjuvant ipilimumab dose #2. Additionally, PBMC from each of the time points will be analyzed for the presence of circulating populations of regulatory T cells, myeloid-derived suppressor cells (MDSC), as well as activated and exhausted T cells.

Tissue Specimens:

•Tumor infiltrating lymphocytes (TILs) will be isolated from the patient's resected tumor and analyzed for infiltrating T cells with specificities against tumor-associated antigens. Additionally, TIL will be analyzed for the presence of infiltrating populations of regulatory T cells, myeloid-derived suppressor cells (MDSC), as well as activated and exhausted T cells.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be in the study if they meet all of the following criteria:

* Histologically or cytologically documented non-small cell lung cancer (NSCLC)
* Clinical stage 1B (≥4cm per CT), Stage 2A/2B, or Stage 3 (N0-2) amenable to surgical resection
* Patients must be deemed a surgical candidate
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* No prior chemotherapy for current diagnosis of lung cancer
* Age is ≥ (greater than or equal to) 18 years
* No active invasive malignancy in the past 2 years other than non-melanoma skin cancer. Cancers that are in-situ are not considered invasive
* Signed written informed consent including Health Insurance Portability and Accountability Act (HIPAA) authorization according to institutional guidelines
* Adequate Organ Function:

  * Absolute neutrophil count (ANC) or absolute granulocyte count (AGC) ≥1500 per microliter (uL)
  * Platelets ≥ 100,000 per uL
  * Total bilirubin ≤(less than or equal to)1.5 milligram per deciliter (mg/dL)
  * Creatinine clearance ≥ 45 milliliter per minute (mL / min); (Creatinine < 2mg / dL to receive cisplatin)
  * Serum glutamic-oxaloacetic transaminase / Serum glutamic pyruvic transaminase (SGOT/SGPT) ≤ 2.5x institutional upper limit normal (ULN)
* Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must test negative for pregnancy within 48 hours prior to any initial study procedure based on a serum pregnancy test. Both sexually active males and females of reproductive potential must agree to use a reliable method of birth control, as determined by the patient and their health care team, during the study and for 3 months following the last dose of study drug. If subject uses appropriate contraceptive methods (the use of two forms at the same time) from the time of the initial serum pregnancy test, then the subsequent pregnancy test can be done within 72 hours of receiving study drug administration. If appropriate contraceptive measures are not begun immediately with the first serum pregnancy test, then subsequent serum pregnancy tests must be done within 48 hours prior to the study drug administration
* Patients must agree to research blood sampling to participate in study

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Have had treatment within the last 30 days with a drug that has not received regulatory (Food and Drug Administration (FDA)) approval for any indication at the time of study entry
* Concurrent administration of any other anti-tumor therapy
* Inability to comply with protocol or study procedures
* Active infection requiring intravenous (IV) antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
* Major surgery (other than definitive lung cancer surgery) within two weeks of study or other serious concomitant systemic disorders that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* Myocardial infarction (MI) having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications
* Contraindication to corticosteroids
* Unwillingness to stop taking herbal supplements while on study
* Female patients who are pregnant or breast-feeding
* Autoimmune disease. Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis)
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* A history of prior treatment with ipilimumab or prior CD137 agonist or cytotoxic T-lymphocyte-associated protein (CTLA 4) inhibitor or agonist
* Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, MD, Principal Investigator — Duke University Medical Center / Thoracic Oncology Program
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Yang CJ, McSherry F, Mayne NR, Wang X, Berry MF, Tong B, Harpole DH Jr, D'Amico TA, Christensen JD, Ready NE, Klapper JA. Surgical Outcomes After Neoadjuvant Chemotherapy and Ipilimumab for Non-Small Cell Lung Cancer. Ann Thorac Surg. 2018 Mar;105(3):924-929. doi: 10.1016/j.athoracsur.2017.09.030. Epub 2017 Dec 16. PMID 29258674

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab: Neoadjuvant: Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes Adjuvant: Ipilimumab 10 mg/kg IV every 3 weeks times 2 doses beginning 4 weeks postoperative ( up to 10 weeks if needed for recovery) Maintenance: Ipilimumab 10 mg/kg/IV every 12 weeks times 2 doses
  Ipilimumab: Neoadjuvant: Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes
  Adjuvant (Post-Surgery): Ipilimumab 10 mg/kg IV every 3 weeks times 2 doses beginning 4 weeks postoperative ( up to 10 weeks if needed for recovery)
  Maintenance: Ipilimumab 10 mg/kg/IV every 12 weeks times 2 doses
  Paclitaxel, Cisplatin, Carboplatin: Neoadjuvant (Pre-Surgery) Cycle 1: Paclitaxel 175 mg/m2 IV over 3 hours , followed by Cisplatin 75 mg/m2 IV over 60 minutes or carboplatin Area Under Curve (AUC) 6 IV over 30-60 minutes on day 1(Every 21 days x 1 cycle)
  Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes, Paclitaxel 175 mg/m2 IV over 3 hours , followed by Cisplatin
Period: Overall Study
Arm/Group | Ipilimumab
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ipilimumab: Neoadjuvant: Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes Adjuvant: Ipilimumab 10 mg/kg IV every 3 weeks times 2 doses beginning 4 weeks postoperative ( up to 10 weeks if needed for recovery) Maintenance: Ipilimumab 10 mg/kg/IV every 12 weeks times 2 doses
  Ipilimumab: Neoadjuvant: Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes
  Adjuvant (Post-Surgery): Ipilimumab 10 mg/kg IV every 3 weeks times 2 doses beginning 4 weeks postoperative ( up to 10 weeks if needed for recovery)
  Maintenance: Ipilimumab 10 mg/kg/IV every 12 weeks times 2 doses
  Paclitaxel, Cisplatin, Carboplatin: Neoadjuvant (Pre-Surgery) Cycle 1: Paclitaxel 175 mg/m2 IV over 3 hours , followed by Cisplatin 75 mg/m2 IV over 60 minutes or carboplatin AUC 6 IV over 30-60 minutes on day 1(Every 21 days x 1 cycle)
  Cycles 2 and 3: Ipilimumab 10 mg/kg IV over 90 minutes, Paclitaxel 175 mg/m2 IV over 3 hours , followed by Cisplatin
Arm/Group | Ipilimumab
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Detectable Circulating T Cells After Treatment
Description: The primary objective of this trial is to determine the percentage of early stage lung cancer patients with detectable circulating T cells specific against tumor-associated antigen (TAA) after receiving platinum based neoadjuvant chemotherapy plus ipilimumab before surgery. Based on Duke intracellular cytokine staining (ICS) assessments over the past 8 years, "detectable" circulating T cells with specificity against TAA are defined as a CD8, CD4, and double positive (DP) (CD4+CD8+) lymphocyte percentage of ≥ 0.05% with each value also being at least twice that of the background unstimulated control value.
Time Frame: 3 months
Population: Intent to treat. Note that the 16.7% of patients that had detectable T-cell responses also had responses at baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 24
Percentage of participants | 16.7

2. Secondary Outcome: Feasibility and Tolerability of Neoadjuvant Chemotherapy Plus Ipilimumab and Surgery
Description: Number of subjects experiencing any of the criteria listed below:
  * Number of subjects receiving 3 doses of preoperative therapy
  * Number of subjects undergoing surgical exploration within 42 days of day 1 of the last cycle of neoadjuvant chemotherapy
  * Number of subjects undergoing lobectomy having surgery-related mortality
  * Number of subjects experiencing dose-limiting toxicity (DLT) during neoadjuvant therapy. DLT will be defined as treatment-related: ≥ Grade 4 hematologic toxicity (excluding neutropenia without fever or infection) or ≥ Grade 3 non-hematologic toxicity (excluding fatigue, nausea, vomiting, peripheral neuropathy, chemotherapy infusion reaction to carboplatin or paclitaxel)
Time Frame: 6 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 24
Participants
  Patients receiving 3 cycles | 24
  Patients undergoing surgical exploration | 13
  Patients undergoing lobectomy | 11
  Patients experiencing a DLT | 3

3. Secondary Outcome: Median Disease-Free Survival
Description: Disease-free survival (DFS) is defined as the time from surgical resection to disease recurrence (first disease recurrence or death, whichever comes first) after surgery. Patients alive who had not recurred as of the last follow-up had DFS censored at the last follow-up date. The Kaplan-Meier estimator will be used to estimate median DFS and its 95% confidence interval.
Time Frame: 5 years
Population: Patients were no longer followed for recurrence following surgery, so this outcome was not captured
Arm/Group | Ipilimumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Subjects Experiencing a Metastasis by Site of Metastasis
Description: Number of patients experiencing a metastasis between baseline and cycle 3
Time Frame: 3 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 24
Participants | 1

5. Secondary Outcome: Patterns of Pathologic Response and Response Evaluation Criteria in Solid Tumor (RECIST) Response
Description: Within each category of RECIST response [partial response (PR), stable disease (SD), progressive disease (PD)], the number of subjects experiencing a pathologic complete response, pathologic partial response, and no pathologic response. RECIST evaluation will be conducted after completion of neoadjuvant therapy. Pathologic response will be evaluated in the resected tumor as follows:
  * No Pathologic Response: No evidence of cell death or tumor necrosis
  * Pathologic Partial Response: ≥30% tumor necrosis or cell death
  * Pathologic Complete Response: No evidence of viable tumor in surgical specimen (includes lung tissue and dissected lymph nodes)
Time Frame: 3 months
Population: Note: pathological response was not captured for study participants. Therefore, the RECIST responses for patients at neoadjuvant month 3 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 24
Participants
  PR | 14
  SD | 8
  PD | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=24)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=24)
Anemia (Blood and lymphatic system disorders) | 21
Atrial fibrillation (Cardiac disorders) | 2
Cardiac disorders - Other, specify: PACS, PATS (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 4
Endocrine disorders - Other, specify: NIGHT SWEATS (Endocrine disorders) | 1
Eye disorders - Other, specify: AURA WHEN READING THIS MORNING (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: GAS (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: GASSY, BURPING (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 4
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 20
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify: FAILURE TO THRIVE (General disorders) | 1
General disorders and administration site conditions - Other, specify: SWEATS X 2 WKS (General disorders) | 1
Infusion related reaction (General disorders) | 2
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 6
Infections and infestations - Other, specify: FOLLICULITIS (Infections and infestations) | 1
Infections and infestations - Other, specify: ORAL CANDIDIASIS (Infections and infestations) | 1
Infections and infestations - Other, specify: PNA ON CXR (Infections and infestations) | 1
Infections and infestations - Other, specify: URI/AUGMENTIN (Infections and infestations) | 1
Infections and infestations - Other, specify: URI/LEVAQUIN (Infections and infestations) | 1
Infections and infestations - Other, specify: UTI ABX X 10 D (Infections and infestations) | 1
Lip infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Creatinine increased (Investigations) | 3
INR increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 10
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: WEAKNESS GENERAL (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Akathisia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 11
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 9
Restlessness (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: GURGLING IN CHEST (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Skin and subcutaneous tissue disorders - Other, specify: DRY CRACKING FINGER NAILS (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: EXCORIATED COCCYX (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: FOLLICULITIS RT DEXAMETHASONE (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: PEELING HANDS/ARMS/FEET/LEGS (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hot flashes (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify: DIAPHORESIS,INTERMITTENT W PAIN (Vascular disorders) | 1
Vascular disorders - Other, specify: VASODILATORY SHOCK (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT01820754/Prot_SAP_000.pdf